CLINICAL TRIAL: NCT06399874
Title: Pilot Trial Comparing Exposure and Nonexposure Treatments for Posttrauma Nightmares and Insomnia: Nightmare Deconstruction and Reprocessing vs. NightWare Wristband
Brief Title: Nightmare Deconstruction and Reprocessing vs. NightWare Wristband
Acronym: NDR/NW
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: NightWare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY-88-13264
Record Dates: First submitted 2024-04-17; First posted 2024-05-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Nightmare
Keywords: Nightmares; Insomnia; PTSD; Heart Rate Variability; Electrodermal Activity; BDNF; Cortisol; ACTH; Treatment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Phase IIa, two-arm, block randomized controlled pilot trial
Who Masked: Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Nightmare Deconstruction and Reprocessing (Experimental): Psychotherapy that uses exposure to nightmare images for trauma activation with the goal of memory reconsolidation.
  Interventions: Behavioral: Nightmare Deconstruction and Reprocessing
- NightWare (Experimental): Wristband device that detects physiologic signals during sleep that indicate a possible nightmare and gently vibrates to rouse the sleeper without fully waking them.
  Interventions: Device: NightWare

INTERVENTIONS:
Behavioral: Nightmare Deconstruction and Reprocessing — A psychotherapy that uses exposure to nightmare images for trauma activation in order to facilitate trauma memory reconsolidation
  Other Names: NDR
  Arms: Nightmare Deconstruction and Reprocessing
Device: NightWare — Wristband device that detects physiologic signals during sleep that indicate a possible nightmare and gently vibrates to rouse the sleeper without fully waking them.
  Other Names: NW
  Arms: NightWare

SUMMARY:
The overall goal of this Phase IIa randomized controlled pilot trial is to assess the potential efficacy of two emerging treatments for post-trauma nightmares and to test the feasibility of study design and methods. Symptom change will be assessed in two treatment arms: (1) Nightmare Deconstruction and Reprocessing (NDR), an exposure-based psychotherapy; and (2) NightWare (NW), a non-exposure approach using a wristband device. The investigators will also assess the feasibility of circadian-dependent blood sampling and use of another wristband to collect physiologic data. Specific aims are: (1) Compare evidence of how well participants tolerate and comply with the two treatments and test feasibility of methods and procedures; (2) Collect additional evidence of the potential efficacy of two contrasting non-pharmacologic approaches to treating posttraumatic nightmares; (3) Explore the operational stress index (OSI) as a reliable, objective measure of sleep disturbance and nightmare events.

DETAILED DESCRIPTION:
This pilot trial is testing two emerging treatments for post-traumatic nightmares: NDR, a novel exposure psychotherapy that targets post-trauma nightmares, and NW, a wristband device that provides non-exposure treatment by detecting physiologic signals of a possible nightmare and gently vibrating to rouse the sleeper without fully waking them. Nightmares and sleep disturbance are important treatment targets because they are prevalent beginning in the acute post-trauma phase and often are long lasting and treatment-resistant. The overall goal of this project is to assess the potential efficacy of these contrasting treatments, which have the potential to treat acute post-trauma nightmares and sleep disturbance in low-resource or far-forward military environments and provide long-term solutions for individuals with treatment-resistant nightmares. The investigators will also test the feasibility collecting biomarker samples at specific time points during treatment, which will provide more information about the potential utility of molecular, neuroendocrine, and physiologic signals of psychological distress related to exposure or non-exposure methods of treating nightmares.

Study Design:

Following up on preliminary studies of NDR and NW, the proposed study will be a Phase IIa, single-blind randomized controlled pilot trial. Up to 30 servicemembers and veterans will be consented. Study duration for each participant is 18 weeks: 6 weeks of observation, 6 weeks of active treatment, and 6 weeks of follow up. Participants have weekly assessments during the observation period, which serves as a within-subjects control. At the end of observation, Participants are randomized to 6 weeks of active treatment in either the NDR or the NW treatment arm. After completing the active treatment period, follow-up assessments are at 2 weeks, 4 weeks, and 6 weeks post-treatment.

Participants in the NW group will receive psychoeducation, equipment instruction, and troubleshooting at each treatment visit. Participants in the NDR group will receive psychoeducation, and NDR treatment at each treatment visit. The investigators will collect blood samples from both treatment groups immediately before and after the first treatment visit (first exposure to nightmares for the NDR arm), and and immediately before and after the final treatment visit (last exposure to nightmares for the NDR arm). All participants will be issued an Empatica EmbracePlus wristband to be worn 23 hours per day. The investigators anticipate that participants in both treatment groups will have a clinically significant decrease in nightmares and nightmare-related sleep disturbance and that molecular, neuroendocrine, and physiologic markers of stress will relate to treatment arm (trauma activation through exposure in NDR or no trauma activation in NW). The investigators also anticipate that biosample collection, processing, and storage methods will be feasible.

Primary and Secondary Outcomes:

The primary outcomes of the proposed trial are nightmare severity and insomnia severity. Nightmare severity will be measured by the Disturbing Dreams and Nightmares Severity Index (DDNSI). Insomnia severity will be assessed using the Insomnia Severity Index (ISI). Nightmare and insomnia severity and variability will be assessed with the DDNSI, the ISI, and EmpaticaPlus wristband data at 14 time points, including screening, once a week during the observation and treatment periods, and follow-up visits.

Secondary outcomes are molecular and neuroendocrine biomarkers (BDNF, cortisol, and ACTH) as well as physiologic parameters (HRV, EDA, and accelerometry data). Change in BDNF, cortisol, and ACTH will be determined through assay of blood samples taken in all treatment groups before and after the first and last treatment sessions. Physiologic data collected via the Empatica EmbracePlus wristband will include HRV and EDA during treatment sessions and accelerometry to track sleep patterns.

ELIGIBILITY:
Inclusion Criteria:

* Active duty service members and veterans
* Minimum symptom severity:
* Has had at least 1 nightmare per week for the past month
* Has a minimum ISI score of 8
* If taking medications for PTSD, depression, anxiety, or insomnia, must be on stable dose for 8 weeks.

Exclusion Criteria:

* Serious risk of suicide
* Psychosis, bipolar disorder, or alcohol or substance use disorder
* Untreated moderate to severe sleep apnea
* Use of synthetic glucocorticoid beta blockers, prazosin, or varenicline
* Current evidence-based or experimental psychotherapy directly targeting nightmares, insomnia, or PTSD
* Inability to recall nightmare content
* Inability to wear wristband or sync wristband data
* Inability to comply with blood draws
* Refusal to consent to DNA analysis of blood samples
* Refusal to consent to audio recording of study visits
* REM sleep behavior disorder or narcolepsy as determined by investigator

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Disturbing Dreams and Nightmare Severity Index | It will be completed at screening, weekly through the observation and treatment periods (12 weeks), and at the 3 follow-up visits (up to 18 weeks post-baseline). It will also be completed at early termination visits, if applicable.
  The DDNSI is a 5-item self-report instrument used to assess nightmare severity and distress both as an inclusion criterion (score ≥10) and as a primary study variable. Possible score range is 0-37, with a recommended cutoff of 10.
Insomnia Severity Index | It will be completed at screening, weekly through the observation and treatment periods (12 weeks), and at the 3 follow-up visits (up to 18 weeks post-baseline). It will also be completed at early termination visits, if applicable.
  The ISI is a 7-item self-report measure that assesses not only perceived severity of insomnia with regards to difficulty falling and staying asleep, but also daytime dysfunction. Possible score range is 0-28, with a recommended cutoff of 8 for sub-threshold insomnia.

SECONDARY OUTCOMES:
Operational Stress Index (OSI) | Collected from baseline through study completion (up to 18 weeks).
  The OSI uses physiological data (heart rate, heart rate variability, skin temperature, movement) to identify stress responses, which may allow researchers to reliably recognize sleep disturbance and nightmare events.
Brain-derived neurotrophic factor (BDNF) levels before and after exposure | Collected at initial NDR exposure component (6 weeks after baseline) and NDR final exposure (12 weeks after baseline).
Cortisol levels before and after exposure | Collected at initial NDR exposure component (6 weeks after baseline) and NDR final exposure (12 weeks after baseline).
Adrenocorticotropic hormone (ACTH) levels before and after exposure | Collected at initial NDR exposure component (6 weeks after baseline) and NDR final exposure (12 weeks after baseline).

CONTACTS AND LOCATIONS:
Overall Officials: James C West, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No